CLINICAL TRIAL: NCT01038895
Title: Aliskiren Versus Ramipril on Antiproteinuric Effect in Hypertensive, Type 2 Diabetic Patients With Microalbuminuria
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Pavia (Other)
Responsible Party: University of Pavia, University of Pavia
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: UNIPV002DIM2009; 2009-016481-83 (Registry Identifier: 2009-016481-83)
Record Dates: First submitted 2009-12-23; First posted 2009-12-24 (Estimated); Last update posted 2009-12-24 (Estimated); Status verified 2009-09

CONDITIONS: Hypertension; Type 2 Diabetes
Keywords: Hypertension; type 2 diabetes; aliskiren; ramipril; microalbuminuria; blood pressure> 130/80 <180/105 mmHg at the end of the wash-out; type 2 diabetes mellitus well controlled by medication and / or; compliance with diet (HbA1c <7%); Microalbuminuria in the upper range of normal (> 200 <300 mg/24 h)
MeSH Terms: conditions — Hypertension; Diabetes Mellitus, Type 2 | interventions — Ramipril

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Ramipril (Active Comparator): 10 mg/daily
  Interventions: Drug: Ramipril
- Aliskiren (Experimental): 300 mg/ daily
  Interventions: Drug: Experimental

INTERVENTIONS:
Drug: Ramipril — tablet; 10 mg; od; 3 months
  Arms: Ramipril
Drug: Experimental — tablet; 300 mg; od; 3 months
  Arms: Aliskiren

SUMMARY:
The main objective of this study is to assess the extent and trend in time of antiproteinuric effect as well as that antihypertensive effect of aliskiren 300 mg / d versus ramipril 10 mg daily in hypertensive patients with type 2 diabetes and microalbuminuria. The investigators will also evaluate:

1. Average of 24 hours, as determined by ABPM, systolic and diastolic blood pressure checks at various visits
2. Average daytime, as determined by ABPM, systolic and diastolic blood pressure checks at various visits 3. Average night, as determined by ABPM, systolic and diastolic blood pressure checks at various visits

ELIGIBILITY:
Inclusion Criteria:

* blood pressure > 130/80 <180/105 mmHg at the end of the wash-out
* type 2 diabetes mellitus well controlled by medication and / or compliance with diet (HbA1c <7%)
* microalbuminuria in the upper range of normal (> 200 <300 mg/24 h)

Exclusion Criteria:

* Pregnancy, lactation or women of childbearing age
* Sitting diastolic blood pressure e 105 mmHg or systolic pressure e 180 at the end of the period of wash-out
* History of hypertensive encephalopathy or cerebrovascular accident within 6 months
* Secondary hypertension
* Heart Failure
* Myocardial infarction within 6 months
* Angina pectoris, clinically significant valvular disease or arrhythmia
* Alteration indices of liver function or renal
* Known hypersensitivity to ACE inhibitors
* All other physiological or pathological condition in the opinion of the physician may affect the evaluation of the parameters under study

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2009-11; Primary Completion 2010-03 (Estimated); Study Completion 2011-06 (Estimated)

PRIMARY OUTCOMES:
Antiproteinuric effect as well as antihypertensive effect of aliskiren 300 mg / daily versus ramipril 10 mg daily in hypertensive patients with type 2 diabetes and microalbuminuria. | 3 months

SECONDARY OUTCOMES:
Average of 24 hours by ABPM, systolic and diastolic blood pressure | 3 months
Average daytime, systolic and diastolic blood pressure | 3 months
Average night, systolic and diastolic blood pressure | 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Roberto Fogari, MD, Study Director — University of Pavia
Locations (1):
- University of Pavia, Pavia, PV, Italy